CLINICAL TRIAL: NCT03126084
Title: Comparison of Postoperative Analgesic Effects of Transversus Abdominis Plane Block and Quadratus Lumborum Block Type 2
Brief Title: Postoperative Effects of TAP Block Versus QLB Type 2 Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANES-QLB-0609
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Inguinal Hernia; Postoperative Pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Acetaminophen; Bupivacaine; Anesthesia, Spinal; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAP (Active Comparator): Patients will undergo inguinal hernia repair under subarachnoid block with 0.5% bupivacaine+glucose.
  Patients will receive transversus abdominis plane block with 20 ml of 0.25% bupivacaine preoperatively, in addition to intravenous acetaminophen 1000mg twice a day for postoperative analgesia.
  Tramadol HCl 50mg intramuscular will be provided for salvage analgesia postoperatively.
  Interventions: Drug: Acetaminophen; Drug: 0.25% Bupivacaine; Drug: 0.5% Bupivacaine+Glucose; Drug: Tramadol HCl; Procedure: Inguinal Hernia Repair
- QLB2 (Active Comparator): Patients will undergo inguinal hernia repair under subarachnoid block with 0.5% bupivacaine+glucose.
  Patients will receive quadratus lumborum type 2 block with 20 ml of %0.25 bupivacaine preoperatively, in addition to intravenous acetaminophen 1000mg twice a day for postoperative analgesia.
  Tramadol HCl 50mg intramuscular will be provided for salvage analgesia postoperatively.
  Interventions: Drug: Acetaminophen; Drug: 0.5% Bupivacaine+Glucose; Drug: Tramadol HCl; Procedure: Inguinal Hernia Repair; Drug: 0.25% Bupivacaine
- CONT (Active Comparator): Patients will undergo inguinal hernia repair under subarachnoid block with 0.5% bupivacaine+glucose.
  Patients will receive intravenous acetaminophen 1000mg twice a day for postoperative analgesia.
  Tramadol HCl 50mg intramuscular will be provided for salvage analgesia postoperatively.
  Interventions: Drug: Acetaminophen; Drug: 0.5% Bupivacaine+Glucose; Drug: Tramadol HCl; Procedure: Inguinal Hernia Repair

INTERVENTIONS:
Drug: Acetaminophen — 1000 mg of intravenous acetaminophen will be administered twice a day
  Other Names: Postoperative routine analgesia
Drug: 0.25% Bupivacaine — 20 ml of 0.25% bupivacaine will be administered to the fascia of the transversus abdominis muscle under ultrasound guidance.
  Other Names: Transversus abdominis plane block
  Arms: TAP
Drug: 0.5% Bupivacaine+Glucose — 15mg of 0.5% bupivacaine will be administered to subarachnoid space through 25G spinal needle
  Other Names: Subarachnoid Block
Drug: Tramadol HCl — 50mg of intramuscular tramadol will be administered when pain score is greater than 3 according to NRS
  Other Names: Postoperative Salvage Analgesia
Procedure: Inguinal Hernia Repair — Patients will undergo open inguinal hernia repair with one of the tension free mesh techniques
Drug: 0.25% Bupivacaine — 10 ml 0.25% bupivacaine will be administered quadratus lumborum muscle and erector spinae muscle
  Other Names: Quadratus lumborum block type 2
  Arms: QLB2

SUMMARY:
This study compares analgesic effectiveness of transversus abdominis plane block and quadratus lumborum block type 2 in open hernia repair surgery. All of the patients will receive routine intravenous analgesic regimen. In addition to that one-third of the patients will receive transversus abdominis plane block, one-third will receive quadratus lumborum block type 2. One-third of the patients will not receive any blocks and will constitute the control group

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 18 years of age
* Patients who are scheduled for elective unilateral open hernia repair with tension free mesh techniques
* Patients who are in ASA's physical status score group 1 or 2

Exclusion Criteria:

* Patients who are younger than 18 years of age
* Patients who have severe stenotic heart diseases
* Patients who have bleeding diathesis
* Patients who have true allergies to local anesthetics
* Patients who have neurologic deficits corresponding to effect site of the anesthetic techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 24 hours after surgery
  Postoperative pain intensity according Numeric Rating Scale between 0-10 (0=no pain, 10=worst pain ever
Pain Intensity | 2 hours after surgery
  Postoperative pain intensity according Numeric Rating Scale between 0-10 (0=no pain, 10=worst pain ever)
Pain Intensity | 6 hours after surgery
  Postoperative pain intensity according Numeric Rating Scale between 0-10 (0=no pain, 10=worst pain ever
Pain Intensity | 48 hours after surgery
  Postoperative pain intensity according Numeric Rating Scale between 0-10 (0=no pain, 10=worst pain ever

CONTACTS AND LOCATIONS:
Overall Officials: Zeki T TEKGUL, MD, Principal Investigator — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Baerentzen F, Maschmann C, Jensen K, Belhage B, Hensler M, Borglum J. Ultrasound-guided nerve block for inguinal hernia repair: a randomized, controlled, double-blind study. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):502-7. doi: 10.1097/AAP.0b013e31825a3c8a. PMID 22705951
- [Background] Finnerty O, Carney J, McDonnell JG. Trunk blocks for abdominal surgery. Anaesthesia. 2010 Apr;65 Suppl 1:76-83. doi: 10.1111/j.1365-2044.2009.06203.x. PMID 20377549
- [Derived] Okur O, Karaduman D, Tekgul ZT, Koroglu N, Yildirim M. Posterior quadratus lumborum versus transversus abdominis plane block for inguinal hernia repair: a prospective randomized controlled study. Braz J Anesthesiol. 2021 Sep-Oct;71(5):505-510. doi: 10.1016/j.bjane.2020.11.004. Epub 2021 Feb 10. PMID 34537121